CLINICAL TRIAL: NCT04241731
Title: A Multicenter Phase II Clinical Study of Cetuximab Plus Raltitrexed for Maintenance Treatment in Advanced Colorectal Cancer
Brief Title: A Study of Cetuximab Plus Raltitrexed for Maintenance Treatment in Advanced Colorectal Cancer
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Jiangsu Cancer Institute & Hospital (Other)
Responsible Party: Principal Investigator, Liangjun Zhu M.M., Ward Director of Internal Medicine, Jiangsu Cancer Institute & Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: JS-GI1901
Record Dates: First submitted 2020-01-23; First posted 2020-01-27 (Actual); Last update posted 2021-08-30 (Actual); Status verified 2021-08

CONDITIONS: Colorectal Cancer
MeSH Terms: conditions — Colorectal Neoplasms | interventions — raltitrexed; Cetuximab

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Raltitrexed Plus Cetuximab (Experimental): Raltitrexed Plus Cetuximab
  Interventions: Drug: Raltitrexed; Drug: Cetuximab

INTERVENTIONS:
Drug: Raltitrexed — Raltitrexed 2.5mg / m2, intravenous infusion for 15min, d1,q2w.
Drug: Cetuximab — Cetuximab 500mg / kg, intravenous drip over 120min, d1,q2w.

SUMMARY:
Maintenance treatment can extend patient survival and improve patient quality of life. Bevacizumab alone or capecitabine combined with bevacizumab as a maintenance treatment have been widely used in clinical practice. In contrast, there are little datas of cetuximab as a maintenance treatment. The purpose of this study is to evaluate efficacy and safety of Raltitrexed plus Cetuximab as the maintenance treatment, and to provide a new choice for RAS wild-type colorectal cancer patients after advanced first-line chemotherapy.

DETAILED DESCRIPTION:
Maintenance treatment can prevent the toxicity and give patients a relative buffer period to alleviate the impact of follow-up treatment on the body without reducing efficacy. Bevacizumab alone or capecitabine combined with bevacizumab as a maintenance treatment have been widely used in clinical practice. There are little datas of cetuximab as a maintenance treatment ,some studies show that Cetuximab is effective in maintenance treatment, and some studies have reported adverse effects of Capecitabine combined with Cetuximab.So it is worthwhile to explore more suitable maintenance treatment options. Raltitrexed, a TS enzyme inhibitor, is an effective chemotherapy drug for colorectal cancer. We plan to evaluate efficacy and safety of Raltitrexed plus Cetuximab in maintenance treatment. Maybe we can provide a new choice for RAS wild-type colorectal cancer patients after advanced first-line chemotherapy.

ELIGIBILITY:
Inclusion Criteria:

* 18-75 years old, no gender restriction;
* RAS wild-type
* Unresectable metastatic colorectal cancer confirmed by histopathology and / or cytology;
* Disease stable or improved while on first-line use of FOLFOX/FOLFIRI with cetuximab for 4-6 months;
* At least one measurable objective tumor lesion by spiral CT scan，the longest diameter measured ≧ 10 mm，or by conventional CT scan，the diameter measured ≧ 20 mm.
* Eastern Cooperative Oncology Group (ECOG) general status score is 0-2;
* Life expectancy of at least 3 months;
* Blood routine, liver and kidney function within the 7 days before screening meet the following criteria: Absolute neutrophil count ≥ 1.5x10^9 / L; hemoglobin ≥ 9.0 g / dl; platelet count ≥ 80 x10^9 / L; total bilirubin ≤ 1.5 times the upper limit of normal (ULN); alanine aminotransferase and aspartate aminotransferase ≤ 2.5 x ULN (≤5 x ULN in patients with liver metastases); ≤3 x ULN in patients with liver metastases (≤5 x ULN in patients with liver metastases); serum creatinine ≤1.5 x ULN;
* Agree to sign informed consent.

Exclusion Criteria:

* BRAF mutant
* Symptomatic brain or meningeal metastases (unless patients receive treatment> 6 months, imaging results are negative within 4 weeks before joining the study, and tumor-related clinical symptoms are stable before joining the study);
* Previous malignant disease within five years, with the exception of the cured primary cervical cancer or basal cell carcinoma of the skin;
* Chronic intestinal disease, infectious intestinal disease, intestinal obstruction, active clinical severe infection and other diseases;
* With ascites
* Substance abuse and medical, psychological or social conditions that may interfere with the participation of patients in the study or influence the evaluation of the results of the study;
* Unsuitable for the study or other chemotherapy determined by investigator.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2019-11-28 (Actual); Primary Completion 2021-11-28 (Estimated); Study Completion 2021-11-28 (Estimated)

PRIMARY OUTCOMES:
The time from the beginning of first-line treatment until the disease progresses. | 24 months
  Progression Free Survival 1.
The time from the beginning of maintenance treatment until the disease progresses. | 24 months
  Progression Free Survival 2.

SECONDARY OUTCOMES:
Overall survival (OS) | 24 months
Incidence of Treatment-Emergent Adverse Events Based on NCI-CTC 4.0 | 24 months
  evaluate the safety of patient medication
Quality of life score | 24 months
  Based on QLQ-C30 in EORTC, evaluate the quality of life of patients

CONTACTS AND LOCATIONS:
Overall Officials: Liangjun Zhu, Study Chair — Jiangsu Cancer Institute & Hospital
Locations (1):
- Jiangsu Cancer Institute & Hospital, Nanjing, Jiangsu, China